CLINICAL TRIAL: NCT01678274
Title: Prospective Characterization of the Heart, Aorta and Blood Pressure in Women With Turner Syndrome. Association With Aortic Dissection.
Brief Title: Prospective Characterization of the Heart, Aorta and Blood Pressure in Turner Syndrome. Association With Aortic Dissection.
Acronym: TSCORII
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 35202
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2015-06

CONDITIONS: Turner Syndrome; Aortic Aneurysm; Ischemic Heart Disease; Hypertension; Congenital Heart Defect
Keywords: Turner Syndrome; Aortic Aneurysm; Ischemic heart disease; Hypertension; Congenital Heart Defect; Pulse Wave Velocity; Augmentation Index; Central Blood Pressure; Agatston Score; Segment involvement score
MeSH Terms: conditions — Turner Syndrome; Aortic Aneurysm; Myocardial Ischemia; Hypertension; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Turner syndrome: Females with Turner syndrome
- Control group: age matched females acting as controls

SUMMARY:
Turner syndrome is a congenital complete or partial lack one of the female sex chromosomes affecting 1 of 2000 live born girls. The syndrome is characterized by an increased prevalence of ischemic heart disease, aortic dilation and dissection, hypertension, stroke and autoimmune diseases in general.

Our study aim is:

* Using MRI to further characterize and find risk factors leading to aortic dilation.
* Using MRI to assess the degree of aortic distensibility.
* Using Computed tomography x-ray scanning of the heart and coronary arteries to characterize the prevalence and degree of ischemic heart disease and coronary anomalies.
* Using pressure sensitive ultrasound (applanation tonometry) to assess the degree of aortic stiffness when compared to controls using end points as Pulse Wave Velocity, Augmentation Index and Central Pulse Pressure.

DETAILED DESCRIPTION:
Turner syndrome is a congenital complete or partial lack one of the female sex chromosomes affecting 1 of 2000 live born girls. The syndrome is characterized by an increased prevalence of ischemic heart disease, aortic dilation and dissection, congenital heart defects, hypertension, stroke, ovarian failure, infertility, decreased final height and autoimmune diseases in general

Our study aim is:

* Using MRI to further characterize and find risk factors leading to aortic dilation.
* Using MRI to describe aortic dimensions
* Using MRI to assess the degree of aortic distensibility.
* Using Computed tomography x-ray scanning of the heart and coronary arteries to characterize the prevalence and degree of ischemic heart disease and coronary anomalies.
* Using pressure sensitive ultrasound (applanation tonometry) to assess the degree of aortic stiffness when compared to controls using end points as Pulse Wave Velocity, Augmentation Index and Central Pulse Pressure.

ELIGIBILITY:
Inclusion Criteria with respect to individuals acting as controls:

* Healthy age matched females

Exclusion Criteria:

* Contraindications for MRI
* Contraindications for CT
* Severe obesity
* Acute og Chronic disease with known or presumed significance with concern to outcomes of the study
* Previous or present malignant disease
* Clinically significant liver disease
* Mechanic or biological heart valves

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females with Turner Syndrome previously participating in our study number 2001024 are recruited from out-patient clinics.
  Controls are healthy volunteers recruited from the general population by advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Aortic dimensions | Once
  Aortic dimensions measured by MRI
Agatston score | Once
  Coronary CT evaluation of Agatston score
Segment involvement score | Once
  Segment involvement score (SIS) calculated as the sum of segments with one or more coronary plaques (score 0-18).
Aortic distensibility | Once
  Aortic distensibillity as measured by MRI

SECONDARY OUTCOMES:
24 hour blood pressure | 24 hour
  24 hour blood pressure
Pulse Wave Velocity | Once
  Pulse Wave Velocity measured by applanation tonometry.
Augmentation index | Once
  Augmentation index measured by applanation tonometry.
Central blood pressure | Once
  Central blood pressure measured by applanation tonometry.

OTHER OUTCOMES:
echocardiography | Once
  echocardiography evaluating Mitral and aortic valves, left ventricular hypertrophy, diastolic and systolic function etc..

CONTACTS AND LOCATIONS:
Overall Officials: Claus H Gravholt, MD, Study Chair — Aarhus University Hospital; Christian Trolle, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Endocrinology and Internal medicine, Aarhus, Denmark

REFERENCES:
- [Derived] Ridder LO, Stochholm K, Mortensen KH, Andersen NH, Gravholt CH. The TGFbeta system and TIMP1 and 3 genotypes in Turner syndrome-Relation with aortic congenital malformations. Clin Endocrinol (Oxf). 2023 Dec;99(6):545-551. doi: 10.1111/cen.14907. Epub 2023 Mar 15. PMID 36890688
- [Derived] Viuff MH, Just J, Brun S, Dam TV, Hansen M, Melgaard L, Hougaard DM, Lappe M, Gravholt CH. Women With Turner Syndrome Are Both Estrogen and Androgen Deficient: The Impact of Hormone Replacement Therapy. J Clin Endocrinol Metab. 2022 Jun 16;107(7):1983-1993. doi: 10.1210/clinem/dgac167. PMID 35302622
- [Derived] Wen J, Trolle C, Viuff MH, Ringgaard S, Laugesen E, Gutmark EJ, Subramaniam DR, Backeljauw P, Gutmark-Little I, Andersen NH, Mortensen KH, Gravholt CH. Impaired aortic distensibility and elevated central blood pressure in Turner Syndrome: a cardiovascular magnetic resonance study. J Cardiovasc Magn Reson. 2018 Dec 13;20(1):80. doi: 10.1186/s12968-018-0497-0. PMID 30541571
- [Derived] Subramaniam DR, Stoddard WA, Mortensen KH, Ringgaard S, Trolle C, Gravholt CH, Gutmark EJ, Mylavarapu G, Backeljauw PF, Gutmark-Little I. Continuous measurement of aortic dimensions in Turner syndrome: a cardiovascular magnetic resonance study. J Cardiovasc Magn Reson. 2017 Feb 24;19(1):20. doi: 10.1186/s12968-017-0336-8. PMID 28231838